CLINICAL TRIAL: NCT02895607
Title: Prospective Evaluation of Outpatient Surgery in the Anterior Cruciate Ligament Reconstructions With Hamstring Hospital
Brief Title: Evaluation of Outpatient Surgery in the Anterior Cruciate Ligament Reconstructions With Hamstring Hospital
Acronym: DIDTGENOU
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: DIDTGENOU
Record Dates: First submitted 2016-09-01; First posted 2016-09-09 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2016-09

CONDITIONS: Anterior Cruciate Ligament

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Ambulatory care among eligible patients — The management of Anterior Cruciate Ligament (ACL) Reconstruction reconstruction in outpatient will be proposed in consultation with the surgeon.
  After an explanation of the course of treatment a fact sheet on the protocol will be provided to the patient and his doctor to the patient to decide its support in CA (ambulatory surgery) or HC (conventional hospitalization).

SUMMARY:
Care in ambulatory surgery (CA) is growing in France, despite lagging behind other countries in North or US Europe. Arthroscopic knee surgery is a minimally invasive surgery eligible for CA. Currently 71.8% of knee arthroscopy are made in this context. However ligamentoplasties anterior cruciate are still carried out predominantly in conventional hospitalization (HC) with a median of 3 to 5.5 days of stay.

Two recent prospective studies French single-operator shows the feasibility of reconstruction of the anterior cruciate ligament (ACL) in ambulatory: no serious events were recorded, the risks are comparable to those of a HC.

However, this support requires a structure and a coordinated network between different medical and paramedical (surgeons, anesthetists, nurse frame, City nurse, doctor, physiotherapist).

The objective of the study is to evaluate (i.e. EPP or "feasibility") ACL reconstruction in CA in hospitals, multi-operator.

DETAILED DESCRIPTION:
II. objectives

at. primary objective

Rating (or "feasibility") of a management protocol HDJ of ACL reconstruction in a hospital structure on a multi-operator series.

Evaluation criteria (absence of EG)?

b. secondary objectives

i. Evaluation of the acceptance rates of ambulatory care patients eligible

ii. Evaluation of the rate and type of complication in our series

iii. Evaluation of early postoperative results (postoperative pain, analgesic consumption, sleep, satisfaction)

IV. Methodology and duration of the research

This is a consecutive series single-center multi-operator prospective regarding the evaluation of surgical practice cited in goal.

The inclusion of patients will take place over a period of 4 months.

The management of ACL reconstruction in outpatient will be proposed in consultation with the surgeon.

After an explanation of the course of treatment a fact sheet on the protocol will be provided to the patient and his doctor to the patient to decide its support AC or HC.

Clinical data will be collected by telephone the first 4 days and in consultation with J45. The revision sheet is provided.

Patients are aware of the use of their data for medical research through oral information provided by the doctor at the signing by the patient's consent related to the surgery.

The data collected as part of the research are anonymous and unidentifiable (for each subject is assigned a number); the name of the surgeon is also anonymized.

ELIGIBILITY:
Inclusion Criteria:

* Isolated ACL tear
* First arthroscopic reconstruction at DIDT

Exclusion Criteria:

* Age over 60 years
* ASA score greater than 2
* Geographical remoteness
* Social isolation
* medical condition requiring supervision by HC (phlebitis history, coagulation disorders ...)
* psychiatric pathology

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients admitted to the orthopedic unit for anterior cruciate ligament (ACL)
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2014-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Assessment of pain by visual analogue scale VAS | Day 45
  Evaluation of pain by visual analogue scale (VAS was numerical scale from 0 = no pain to 10 = unbearable pain)

SECONDARY OUTCOMES:
Assessment of sleep quality | Day 45
  Quality sleep (ENS = 0 = 10 complete insomnia deep sleep without interruption)
Assessment of Patient satisfaction | Day 45
  Patient satisfaction (ENS 0 = very dissatisfied to 10 = very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Emmanuel MOREAU, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided